CLINICAL TRIAL: NCT05588414
Title: Performance Assessment of the Fluorescence Technique Alone in the Search for the Sentinel Node in Breast Surgery, Compared to the Use of the Combined Fluorescence and Isotopic Method
Brief Title: Performance Assessment of the Fluorescence Technique Alone in the Search for the Sentinel Node in Breast Surgery
Acronym: FLUORES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-04
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green fluorescence method as first step (Other): Systematic double identification of the sentinel lymph node, by sequential use of ICG fluorescence technique as first step followed by isotopic technique.
  Interventions: Procedure: Standardization of the sentinel node detection procedure

INTERVENTIONS:
Procedure: Standardization of the sentinel node detection procedure — All patients included in the study underwent the same pre- and intra-operative procedure, consisting of a double systematic sentinel node detection, using sequential ICG and isotopic technique. The patient is his own control for the analysis of the performance of the ICG technique alone compared to the combined ICG and isotopic technique.

SUMMARY:
Cohort, interventional, multicenter, non-randomized study to compare the performance of the ICG fluorescence technique (ICG) alone to the combined ICG + isotopic technique in the detection of sentinel node.

Comparison of the performances of two techniques used in current practice, without modification of the patients' care plan. Indeed, all patients receive both techniques, but the protocol allows to standardize the collection of the performances of each of the two techniques in order to compare them.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age on the day of inclusion,
* Presenting with breast cancer,
* Fulfilling the Sentinel Node search criteria of:

  * Patient with carcinoma in situ with high risk of microinvasion:
* nodular presentation, high grade with necrosis,
* suspicion of microinvasion at biopsy,
* radiological size of more than 40 mm,
* need for mastectomy or extensive resection requiring a complex oncoplasty surgery (no size criteria, at the surgeon's discretion)

  * Patient with T1-T2 invasive carcinoma AND no lymph node involvement according to Tumor-Node-Metastasis (TNM) classification (N0) on clinical and imaging (negative axillary echo or negative lymph node biopsy):
* unifocal or bifocal proximal tumor
* < 5 cm (clinical), palpable or non-palpable (subcentimetric allowed)
* in case of neoadjuvant chemotherapy: before or after if N0 and negative axillary echo or negative biopsy
* Benefiting from a French social security system
* Having been informed of the study and having freely given their informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Patient not eligible for the sentinel node procedure (contraindication to surgery, N+ and/or M+ clinical or radiological, T3 and more, history of homolateral breast cancer surgery)
* Patient under guardianship or curators
* Patient under court protection
* Patient who does not understand French
* Patient already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (Sensitivity and Specificity) of the indocyanine green fluorescence (ICG) method | At time of surgery
  The main objective is to evaluate the diagnostic performance (Sensitivity and Specificity) of the indocyanine green fluorescence (ICG) method alone as a sentinel node marker in non-metastatic breast cancer, compared to the method coupling technetium-99m isotopic research (TC) to fluorescence (Gold Standard in the study centers).
  The suspicious node bundles, which will have been removed after identification by 1) ICG alone, 2) TC alone or 3) manually, can be classified in a contingency table, according to the first method (the sequence) with which they are detected.
  The Sensitivity / Specificity pair will then be used to :
  1. Estimate the area under the curve (AUC) of the ICG method alone, and its 95% confidence interval.
  2. Estimate the positive and negative predictive values of ICG alone, using the prevalence of metastatic lesions.

SECONDARY OUTCOMES:
Frequency and factors associated with the occurrence of false negatives (FN) related to the use of ICG alone (fluorescence tracking failure alone) | At time of surgery
  The number and percentage of lymph node packages detected only by isotopic method. Analysis of the factors (patient characteristics such as total mastectomy vs. partial mastectomy, obesity, tumor location in the mammary gland) associated with the occurrence of these false negatives, using a multivariate logistic regression model.
Frequency of detection on table by multispectral camera, of ganglions first detected only by isotopic method. | At time of surgery
  Number and percentage of ganglion bundles detected only by isotopic method, among which we will finally find a marking with the multispectral camera.
Causes of premature use of the isotope method (moving to the second stage of tracking) before the first stage of tracking (ICG method) has been completed. | At time of surgery
  Frequencies of pre-identified causes of premature isotopic use during the first stage of the axillary procedure. The pre-identified causes are the follows:
  * Poor skin visualization
  * Operative difficulty with persistence of a fluorescent signal
  * Loss of fluorescent signal
  * Loss of surgeon patience
  * Other.
Surgeon's perception of the usefulness and self-perceived satisfaction of ICG method alone, compared with the combined technique (ICG+TC). | At time of surgery
  Description of the surgeon's self-perceived satisfaction with the use of the ICG alone, using individualized 10-point Likert scales (0 = not at all useful/satisfied; 10 = quite useful/satisfied).
Interest of the ICG technique alone compared to the combined technique for the detection of metastases. | Upon receipt of the anatomopathology results
  Diagnostic performance of ICG method to identify sentinel node will be associated with the frequency of detection of metastases (weighted by the number of nodes present in the lymph node packages sent to pathology) in order to evaluate the diagnostic performance of this method as sentinel metastatic node marker.

CONTACTS AND LOCATIONS:
Overall Officials: Didier TARDIF, Doctor, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (5):
- France (5):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Hôpital Privé Drôme Ardèche, Guilherand-Granges
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No